CLINICAL TRIAL: NCT00104052
Title: Assessment of the Safety, Efficacy, Tolerability and Pharmacokinetics of PEG-Intron® Plus REBETOL® in Pediatric Patients With Chronic Hepatitis C
Brief Title: Study of PEG-Intron Plus REBETOL in Pediatric Subjects With Chronic Hepatitis C (Study P02538 Part 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02538: Part 1
Record Dates: First submitted 2005-02-22; First posted 2005-02-23 (Estimated); Results first posted 2009-03-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-Intron alfa 2b (PEG2b) plus REBETOL (RBV) (Experimental): PEG2b 1.5 μg/kg/wk given subcutaneously (once weekly) and RBV 400-1200 mg/day by mouth divided in 2 daily doses (administered twice daily with food, dosed 12 hours apart) for 48 weeks. Subjects treated up to 48 weeks and followed for additional 24 weeks after the end of treatment (total of 72 weeks study participation).
  Interventions: Biological: peginterferon alfa-2b (PEG2b) (SCH 54031); Drug: ribavirin (SCH 18908)

INTERVENTIONS:
Biological: peginterferon alfa-2b (PEG2b) (SCH 54031) — PEG2b 1.5 μg/kg/wk given subcutaneously (once weekly) for 48 weeks.
  Other Names: PEG-Intron (SCH 54031)
Drug: ribavirin (SCH 18908) — 15 mg/kg/day for up to 48 weeks
  Other Names: REBETOL (SCH 18908)

SUMMARY:
The primary objective is to assess the safety, efficacy and tolerability of the combination of PEG-Intron plus REBETOL in pediatric subjects with chronic hepatitis C. The secondary objective is to measure the multiple-dose pharmacokinetics of PEG-Intron and REBETOL in pediatric subjects with chronic hepatitis C.

DETAILED DESCRIPTION:
This global, multicenter, open-label Phase 3 study will evaluate the safety, efficacy and tolerability of PEG-Intron plus REBETOL in previously untreated pediatric subjects, ages 3 through 17 years, with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3-17 years old
* Individuals weighing ≤ 90 kg
* Previously untreated children with chronic hepatitis C (HCV RNA qPCR plasma positive)
* Individuals with any HCV (hepatitis C virus) genotype
* Hematology laboratory results of:

  * Hemoglobin (HGB) ≥ 11 g/dL for females or ≥ 12g/dL for males,
  * White Blood Cell Count (WBC) ≥ 3,000/mm^3,
  * Neutrophils ≥ 1,500/mm^3,
  * Platelets ≥ 100,000/mm^3
* Chemistry laboratory results of:

  * Normal Thyroid Stimulating Hormone (TSH), albumin, creatinine, and Bilirubin,
  * Antinuclear antibody (ANA) ≤ 1:160,
  * Fasting Glucose 70-140 mg/dL. Note: If glucose levels are between 116-140 mg/dL or an individual has diabetes, HbA1C must be ≤ 8.5%
* Compensated liver disease
* Historic or pre-treatment liver biopsy slides available
* No significant co-existing psychiatric disease
* Those with diabetes, hypertension, or birth prior to 32 weeks gestational age must have normal eye exams and retinal photographs (these will be done as part of the study before hepatitis C treatment is given)
* Patients and partners of patients willing to use adequate contraception during the course of the study
* Abstain from alcohol and any other illicit drugs

Exclusion Criteria:

* Serum ALT >10 times the upper limit of normal within the 6 months prior to study
* Previous hepatitis C treatment
* Children with liver disease not caused by hepatitis C
* Most recent liver biopsy is normal
* Individuals infected with the hepatitis B virus and/or human immunodeficiency virus (HIV)
* Known blood disorders such as hemoglobinopathy, coagulopathy, or G6PD deficiency
* Known immunodeficiency disorders requiring immunoglobulin therapy
* Body organ transplant
* Any known or suspected cancer within the past 5 years
* Children with chronic pulmonary disease
* Individuals who have a medical condition that would likely require systemic steroids
* Those with a history of central nervous system (CNS) trauma or seizure disorders
* Individuals with pre-existing psychiatric disorders including but not limited to moderate to severe depression
* Current or previous use of lithium or antipsychotic drugs
* Patients with clinically significant electrocardiogram (ECG) abnormalities and/or significant cardiovascular dysfunction (e.g., angina, congestive heart failure, recent myocardial infarction, uncontrolled hypertension, significant arrhythmia, cardiac sequelae from Kawasaki disease, cardiomyopathy, and/or history of congenital heart disease)
* Insulin-dependent diabetes mellitus or poorly controlled non-insulin dependent diabetes mellitus
* Immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, or symptomatic thyroid disorder)
* History of substance abuse, including alcohol (e.g., binge drinking, blackouts), intravenous drugs and inhaled drugs
* Subjects who have a history of pregnancy or who are pregnant and/or breast feeding. Subjects who intend to become pregnant during the study period. Subjects with partners who intend to become pregnant during the study period
* Subjects with clinically significant retinal abnormalities such as known retinopathy of prematurity or other retinopathies

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2005-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Haber B, Alonso E, Pedreira A, Rodriguez-Baez N, Ciocca M, Lacaille F, Lang T, Gonzalez T, Goodman Z, Yang Z, Jackson B, Noviello S, Albrecht JK. Long-Term Follow-Up of Children Treated With Peginterferon and Ribavirin for Hepatitis C Virus Infection. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):89-94. doi: 10.1097/MPG.0000000000001239. PMID 27111344
- [Derived] Wirth S, Ribes-Koninckx C, Calzado MA, Bortolotti F, Zancan L, Jara P, Shelton M, Kerkar N, Galoppo M, Pedreira A, Rodriguez-Baez N, Ciocca M, Lachaux A, Lacaille F, Lang T, Kullmer U, Huber WD, Gonzalez T, Pollack H, Alonso E, Broue P, Ramakrishna J, Neigut D, Valle-Segarra AD, Hunter B, Goodman Z, Xu CR, Zheng H, Noviello S, Sniukiene V, Brass C, Albrecht JK. High sustained virologic response rates in children with chronic hepatitis C receiving peginterferon alfa-2b plus ribavirin. J Hepatol. 2010 Apr;52(4):501-7. doi: 10.1016/j.jhep.2010.01.016. Epub 2010 Feb 4. PMID 20189674

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-Intron Plus REBETOL: SCH 54031 PEG-Intron (peginterferon alfa-2b) 60 µg/m2 subcutaneous injection once weekly plus SCH 18908 REBETOL (ribavirin) 15 mg/kg PO daily in two divided doses for 48 weeks for subjects with Genotypes 1,4,5,6 and high-viral-load (≥600,000 IU/mL) Genotype 3 subjects. For subjects with Genotype 2 or low-viral-load Genotype 3 (<600,000 IU/mL), the same treatment will be given for 24 weeks.
Period: Overall Study
Arm/Group | PEG-Intron Plus REBETOL
Started | 107
Completed | 78
Not Completed | 29
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 26
Not completed — Discontinuation unrelated to treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | PEG-Intron Plus REBETOL
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Virologic Response (SVR) at 24 Weeks Post-treatment
Description: SVR is defined as undetectable hepatitis C virus ribonucleic acid (HCV-RNA) at 24 weeks post-treatment
Time Frame: Up to 48-week treatment duration. Follow-up of 24 weeks.
Population: Carry Forward analysis of participants who received at least one dose of study medication. This dataset includes one subject with undetectable HCV-RNA at Follow-up Week 12 (FW 12) but missing data at FW 24; this subject was considered a sustained responder in the Carry Forward analysis.
Measure: Number; unit: Participants
Arm/Group | PEG-Intron Plus REBETOL
Number analyzed (Participants) | 107
Participants | 70
Statistical Analysis 1: Comparison: PEG-Intron Plus REBETOL; Test type: Superiority or Other; Normal approximation to the binomial = 0.654, 95% CI [0.564 to 0.744]

ADVERSE EVENTS:
Arm/Group | PEG-Intron Plus REBETOL
Serious Adverse Events (participants affected / at risk) | 3/107
Other Adverse Events (participants affected / at risk) | 107/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron Plus REBETOL (N=107)
PALPITATIONS (Cardiac disorders) | 1 (1)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron Plus REBETOL (N=107)
ANAEMIA (Blood and lymphatic system disorders) | 12 (20)
LEUKOPENIA (Blood and lymphatic system disorders) | 11 (15)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 10 (14)
NEUTROPENIA (Blood and lymphatic system disorders) | 35 (61)
EYE PAIN (Eye disorders) | 6 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 28 (58)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 (24)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 6 (12)
DIARRHOEA (Gastrointestinal disorders) | 16 (20)
NAUSEA (Gastrointestinal disorders) | 22 (41)
VOMITING (Gastrointestinal disorders) | 36 (76)
ASTHENIA (General disorders) | 16 (40)
CHILLS (General disorders) | 23 (58)
FATIGUE (General disorders) | 32 (125)
INFLUENZA LIKE ILLNESS (General disorders) | 10 (51)
INJECTION SITE ERYTHEMA (General disorders) | 31 (50)
IRRITABILITY (General disorders) | 16 (42)
MALAISE (General disorders) | 10 (24)
PAIN (General disorders) | 10 (20)
PYREXIA (General disorders) | 86 (617)
NASOPHARYNGITIS (Infections and infestations) | 11 (15)
PHARYNGITIS (Infections and infestations) | 6 (7)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 6 (6)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 6 (9)
WEIGHT DECREASED (Investigations) | 20 (29)
ANOREXIA (Metabolism and nutrition disorders) | 31 (41)
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 (34)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 (70)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (13)
MYALGIA (Musculoskeletal and connective tissue disorders) | 20 (100)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (28)
DIZZINESS (Nervous system disorders) | 15 (25)
HEADACHE (Nervous system disorders) | 71 (410)
NERVOUSNESS (Psychiatric disorders) | 9 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 24 (31)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (10)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 15 (20)
ACNE (Skin and subcutaneous tissue disorders) | 6 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 19 (21)
DRY SKIN (Skin and subcutaneous tissue disorders) | 15 (19)
ECZEMA (Skin and subcutaneous tissue disorders) | 9 (11)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 8 (9)
RASH (Skin and subcutaneous tissue disorders) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less